CLINICAL TRIAL: NCT04193631
Title: A Controlled-Dose Study Using A One Time Low Dose Cannabidiol Tablet For The Treatment of Mild to Moderate Musculoskeletal Pain
Brief Title: Low Dose of Cannabidiol (CBD) to Treat Mild to Moderate Musculoskeletal Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pure Green (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-19-00A
Record Dates: First submitted 2019-12-08; First posted 2019-12-10 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Musculoskeletal Pain
Keywords: CBD; Cannabidiol; Musculoskeletal Pain; Pain
MeSH Terms: conditions — Musculoskeletal Pain; Pain | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pure Green Tablet (Experimental): A water-soluble sublingual tablet that contains 5 mg of cannabidiol (CBD).
  Interventions: Drug: Cannabidiol (CBD)

INTERVENTIONS:
Drug: Cannabidiol (CBD) — A single dose of Cannabidiol (CBD) when patients experience musculoskeletal pain in the trial.

SUMMARY:
The purpose of the study is to evaluate whether Pure Green tablets is a better pain reliever for the treatment of mild to moderate musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 21 years of age;
2. Subject has mild to moderate musculoskeletal pain;
3. Pain for greater than or equal to 10 days of each month for 3 months prior to study entry for which the pain requires treatment.
4. Has an Numeric Pain Rating Scale (NPRS) score of 3 or greater,
5. If female, subject is practicing an approved method of birth control throughout the study;
6. Subject is willing and able to comply with all protocol-specified requirements;
7. Subject is willing to take Pure Green tablets only and will not take any other pain medications,
8. Subject is willing to provide his/her written informed consent to participate in the study as stated in the informed consent document.
9. Subject is willing to document pain scale scores in a diary.

Exclusion Criteria:

1. Subject has any condition for which the investigator does not feel the participant should be enrolled due to possible safety or compliance issues;
2. Subject has received treatment with an investigational drug or therapy within 30 days or 5 half-lives (whichever is longer) prior to Day 1.
3. Subject has a known allergy to active or inert ingredients of Pure Green tablets;
4. Subject is taking a concomitant medication or treatment that would complicate use or interpretation of the study drug's effects (examples include: Cannabis (marijuana) or any cannabinoid products including Cannabidiol (CBD) or Tetrahydrocannabinol (THC); Any drug or herbal product that influences the endocannabinoid system (ECS));
5. Have serious cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
6. Have a history of recurrent seizures other than febrile seizures.
7. Have current or pending disability compensation or litigation issues that may compromise response to treatment, in the opinion of the investigator.
8. Have a diagnosis of inflammatory arthritis (that is, rheumatoid arthritis) or an autoimmune disorder (excluding inactive Hashimoto's thyroiditis).
9. Use of acupuncture, chiropractic maneuvers, transcutaneous electrical nerve stimulation (TENS), or similar procedures aimed to relieve any kind of pain.
10. Patients who are anticipated by the investigator to require use of analgesic agents including but not limited to non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen/paracetamol, and opioids, or other excluded medication for the duration of the study.
11. Are unwilling or unable to comply with the data collection method used to record their patient rated outcome data.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Impact of Pure Cannabidiol (CBD) tablets on safety in patient's with musculoskeletal pain using a self-reported pain scale score. | 1 Day
  To evaluate the safety and efficacy of Pure Green Cannabidiol (CBD) sublingual tablets for the treatment of musculoskeletal pain by having patients evaluate their Numeric Pain Rating Scale (NPRS) score reported as 0-10 where 0 is no pain and 10 is the worst pain possible.

SECONDARY OUTCOMES:
To evaluate efficacy of a low dose of Cannabidiol (CBD) in the treatment of mild to moderate musculoskeletal pain. | 1 Day
  To explore the impact of Pure Green sublingual tablets on patient self-reported Numeric Pain Rating Scale (NPRS), as a route of administration and reduction in baseline pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kimless, MD, Principal Investigator — Chief Medical Officer
Locations (1):
- Dr. Kimless' Clinic, Chadds Ford, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madden K, van der Hoek N, Chona S, George A, Dalchand T, Baldawi H, Mammen G, Bhandari M. Cannabinoids in the Management of Musculoskeletal Pain: A Critical Review of the Evidence. JBJS Rev. 2018 May;6(5):e7. doi: 10.2106/JBJS.RVW.17.00153. No abstract available. PMID 29787450
- [Background] Hill KP, Palastro MD, Johnson B, Ditre JW. Cannabis and Pain: A Clinical Review. Cannabis Cannabinoid Res. 2017 May 1;2(1):96-104. doi: 10.1089/can.2017.0017. eCollection 2017. PMID 28861509
- [Background] Therapeutic Effects of Cannabis and Cannabinoids, National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Population Health and Public Health Practice; Committee on the Health Effects of Marijuana: An Evidence Review and Research Agenda. Washington (DC): National Academies Press (US); 2017 Jan 12.
- [Background] Ware MA, Wang T, Shapiro S, Collet JP; COMPASS study team. Cannabis for the Management of Pain: Assessment of Safety Study (COMPASS). J Pain. 2015 Dec;16(12):1233-1242. doi: 10.1016/j.jpain.2015.07.014. Epub 2015 Sep 16. PMID 26385201